CLINICAL TRIAL: NCT00522106
Title: The Effectiveness of Behavioral Graded Activity in Patients With Osteoarthritis of the Hip and/or Knee: a Randomized Controlled Trial
Brief Title: The Effectiveness of Behavioral Graded Activity in Patients With Osteoarthritis of the Hip and/or Knee
Acronym: GRADIT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Netherlands Instititute for Health Services Research (Other)
Collaborators: Amsterdam UMC, location VUmc (Other); UMC Utrecht (Other); Maastricht University (Other); Radboud University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GRADIT-01
Record Dates: First submitted 2007-08-28; First posted 2007-08-29 (Estimated); Last update posted 2007-08-29 (Estimated); Status verified 2007-08

CONDITIONS: Osteoarthritis
Keywords: Behavioral graded activity; Hip; Knee; Physical therapy; Exercise therapy
MeSH Terms: conditions — Osteoarthritis | interventions — Exercise Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Behavioral graded activity
  Interventions: Behavioral: Behavioral graded activity
- B (Active Comparator): Exercise therapy
  Interventions: Other: Exercise therapy

INTERVENTIONS:
Behavioral: Behavioral graded activity — The intervention is directed at increasing the level of activities in a time-contingent way, with the goal to integrate these activities in the daily living of the patients. The intervention is performed by physical therapists in primary care, on individual basis. Treatment period of maximal 12 weeks (with maximal 18 sessions), followed by 5 pre-set boostermoments with a maximum of 7 sessions (respectively in week 18, 25, 34, 42, and 55).
  Arms: A
Other: Exercise therapy — Treatment according to the Dutch physiotherapy guideline for patients with osteoarthritis of hip and/or knee. This guideline consists of general recommendations, emphasizing provision of information and advice, exercise therapy, and encouragement of a positive coping with the complaints. The treatment consisted of a maximum of 18 sessions within a period of 12 weeks. The treatment could be discontinued within the 12 week period if, according to the physiotherapists, all treatment goals were achieved.
  Arms: B

SUMMARY:
We performed a randomized controlled trial to study the effectiveness of Behavioral graded activity (BGA) in patients with OA of the hip or knee. It was hypothesised that in the long term BGA results in less pain, less limitations in activities, and better patient global assessment (i.e. the effect of treatment perceived by patients themselves), compared to usual care of physiotherapists (UC). UC was operationalized as physiotherapeutic care according to the Dutch physiotherapy guideline for patients with hip and/or knee OA. It was also investigated whether specific subgroups of patients benefited more from BGA and which factors influenced the success of BGA-treatment. Also, it will be investigated whether differences exist in exercise adherence and whether there is a relationship between exercise adherence and long-term effectiveness.

DETAILED DESCRIPTION:
The principle objectives of managing OA are to control pain adequately, improve function and reduce disability. There is strong evidence that exercise therapy has a short term benefit for OA. However, these beneficial effects decrease over time and finally disappear. This decline is thought to be related to the difficulties people have in maintaining adherence to prescribed exercises. Therefore, to enhance long term benefit, adherence to exercise therapy is of utmost importance. Recently, the focus of attention within physiotherapy has shifted towards behaviorally oriented treatment, like Behavioral Graded Activity (BGA), which focuses less on pain and includes psychological and social factors in the treatment-process. Such intervention seems appropriate to increase the level of activities of patients with OA in a time-contingent way and to increase patients' adherence to these activities.

However, at the start of the present study the scientific evidence for the effectiveness of BGA in patients with a progressive and specific chronic disease, like OA of the hip and knee, was not available. Therefore, we performed a randomized controlled trial to study the effectiveness of BGA in patients with OA of the hip or knee. It was hypothesised that in the long term BGA results in less pain, less limitations in activities, and better patient global assessment (i.e. the effect of treatment perceived by patients themselves), compared to usual care of physiotherapists (UC). UC was operationalized as physiotherapeutic care according to the Dutch physiotherapy guideline for patients with hip and/or knee OA. It was also investigated whether specific subgroups of patients benefited more from BGA and which factors influenced the success of BGA-treatment. Also, it will be investigated whether differences exist in exercise adherence and whether there is a relationship between exercise adherence and long-term effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Osteoarthritis of hip or knee according to the clinical criteria of the American College of Rheumatology

Exclusion Criteria:

* other pathology explaining the complaints;
* complaints in less than 10 out of 30 days;
* treatment for these complaints with exercise therapy in the preceding six months;
* under 50 or over 80 years of age;
* indication for hip or knee replacement within one year;
* contraindication for exercise therapy;
* inability to understand the Dutch language;
* a high level of physical function (since patients who perform at a high level of physical function at baseline do not need to increase their level of physical function. A high level of physical function was operationalized on a score of less than two on the sections walking ability and physical function of the Algofunctional index)

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2001-05; Study Completion 2008-05 (Estimated)

PRIMARY OUTCOMES:
Pain | week 0, 13, 39 and 65
Physical function | week 0, 13, 39 and 65
Patient global assessment | week 13, 39 and 65

SECONDARY OUTCOMES:
Tiredness | week 0, 13, 39 and 65
Stiffness | week 0, 13, 39 and 65
Joint mobility | week 0, 13, and 65
Muscle strength | week 0, 13, and 65
Patient-specific physical function | week 0, 13, 39 and 65
Walking test | week 0, 13, and 65
Pain coping | week 0, and 65
Locus of control | week 0 and 65
Quality of life | week 0, 13, 39 and 65
Exercise adherence | week 13, 39 and 65
Social support | week 0, and 65
Level of performed activities | week 0, 13, 39 and 65

CONTACTS AND LOCATIONS:
Overall Officials: Joost Dekker, PhD, Study Director — VU Medical Center Amsterdam, The Netherlands; Johannes WJ Bijlsma, PhD, MD, Study Director — UMC Utrecht, The Netherlands; Cindy Veenhof, PhD, Principal Investigator — NIVEL, Utrecht, The Netherlands; Cornelia HM van den Ende, PhD, Study Director — St Maartenskliniek, Nijmegen, The Netherlands; Martijn FP Pisters, MSc, Principal Investigator — NIVEL, Utrecht, The Netherlands
Locations (1):
- NIVEL, Utrecht, Netherlands

REFERENCES:
- [Result] Veenhof C, Koke AJ, Dekker J, Oostendorp RA, Bijlsma JW, van Tulder MW, van den Ende CH. Effectiveness of behavioral graded activity in patients with osteoarthritis of the hip and/or knee: A randomized clinical trial. Arthritis Rheum. 2006 Dec 15;55(6):925-34. doi: 10.1002/art.22341. PMID 17139639
- [Result] Veenhof C, van Hasselt TJ, Koke AJ, Dekker J, Bijlsma JW, van den Ende CH. Active involvement and long-term goals influence long-term adherence to behavioural graded activity in patients with osteoarthritis: a qualitative study. Aust J Physiother. 2006;52(4):273-8. doi: 10.1016/s0004-9514(06)70007-1. PMID 17132122
- [Result] Coupe VM, Veenhof C, van Tulder MW, Dekker J, Bijlsma JW, Van den Ende CH. The cost effectiveness of behavioural graded activity in patients with osteoarthritis of hip and/or knee. Ann Rheum Dis. 2007 Feb;66(2):215-21. doi: 10.1136/ard.2006.054478. Epub 2006 Jul 31. PMID 16880195
- [Result] Veenhof C, Dekker J, Bijlsma JW, van den Ende CH. Influence of various recruitment strategies on the study population and outcome of a randomized controlled trial involving patients with osteoarthritis of the hip or knee. Arthritis Rheum. 2005 Jun 15;53(3):375-82. doi: 10.1002/art.21171. PMID 15934129
- [Derived] Pisters MF, Veenhof C, de Bakker DH, Schellevis FG, Dekker J. Behavioural graded activity results in better exercise adherence and more physical activity than usual care in people with osteoarthritis: a cluster-randomised trial. J Physiother. 2010;56(1):41-7. doi: 10.1016/s1836-9553(10)70053-9. PMID 20500136
- [Derived] Pisters MF, Veenhof C, Schellevis FG, De Bakker DH, Dekker J. Long-term effectiveness of exercise therapy in patients with osteoarthritis of the hip or knee: a randomized controlled trial comparing two different physical therapy interventions. Osteoarthritis Cartilage. 2010 Aug;18(8):1019-26. doi: 10.1016/j.joca.2010.05.008. Epub 2010 May 19. PMID 20488250